CLINICAL TRIAL: NCT03306004
Title: Neonatal Jaundice: Knowledge, Attitudes and Practices of Mothers and Medical Trainees and Providers in and Around Ogbomosho
Acronym: 4NNJ
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HSR 16_2172x
Record Dates: First submitted 2017-09-01; First posted 2017-10-10 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Health Care Providers: Providers answer questionaires
  Interventions: Other: Questionare
- Mothers: Mothers answer questionaires
  Interventions: Other: Questionare

INTERVENTIONS:
Other: Questionare

SUMMARY:
Determine the knowledge attitude and practices of all levels of health care providers about neonatal jaundice

DETAILED DESCRIPTION:
During the routine post-natal visit, trained research personnel will inform the mother of the infant or medical practitioner that a study in being carried out to better understand the knowledge, attitudes and practices of mothers and health care providers for neonatal jaundice. The investigators will then proceed to ask the mothers or health care professionals if they would be interested in filling out an anonymous survey that will assess their knowledge of neonatal jaundice and their practices, if any, in caring for this condition. No PHI will be included and no written consent will be obtained as the written consent would be the only link to the person participating in the survey. Verbal consent will be obtained and we will explain that their medical care and care of the children will in no way be affected by their answers to the survey. We will carefully explain that their participation in the survey is voluntary.

For medical students, they will be informed that a study is being carried out to better understand the knowledge, attitudes and practices of medical trainees for neonatal jaundice. They will then be asked if they would be interested in filling out an anonymous survey that assess their knowledge of neonatal jaundice, and their practices, if any, in caring for this condition. No PHI will be included and no written consent will be obtained, as the written consent would be the only link to the person participating in the survey. Verbal consent will be obtained and we will explain that their academic standing will not be affected by their answers to the survey. We will carefully explain that their participation in the survey is voluntary.

All surveys will contain the names and contact information of the investigators.

The survey will be administered under the direction of the researchers by the researchers and/or their trained research team.

ELIGIBILITY:
Inclusion Criteria:

* All Mothers and Health Care Workers willing to fill out survey in and around Ogbomoso, Nigeria

Exclusion Criteria:

* All Mothers and Health Care Workers not willing to fill out survey in an around Ogbomoso, Nigeria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health Care providers and Mothers with neonates in for routine childcare visits
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Knowledge of Jaundice | Baseline
  Assess the knowledge of health care and mothers regarding jaundice in neonates using a multi choice survey with approximately 40 questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Bowen University Teaching Hospital, Ogbomoso, Nigeria

IPD SHARING:
Plan to Share IPD: No